CLINICAL TRIAL: NCT02270866
Title: Effects of Neuromodulation on Verbal Fluency in Post-stroke Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scion NeuroStim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: SNS-APH-01
Record Dates: First submitted 2014-10-14; First posted 2014-10-21 (Estimated); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Post-stroke Aphasia
Keywords: aphasia; stroke
MeSH Terms: conditions — Aphasia; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Caloric Vestibular Stimulation (CVS) (Experimental)
  Interventions: Device: TNM Device

INTERVENTIONS:
Device: TNM Device — The device is worn like a music headset and the patient lies on a wedge pillow while the device is active. Each session lasts under 20 minutes.

SUMMARY:
This is a single site, open label study with a single arm designed to assess the feasibility of use of caloric vestibular stimulation (CVS) in patients with post-stroke aphasia. CVS is delivered via a portable, non-invasive device. Both language and movement assessments are made.

ELIGIBILITY:
Inclusion Criteria:

* >6 months post-stroke (ischemic or hemorrhagic)
* receptive or expressive aphasia
* little or no improvement in language ability in the preceding 3 months

Exclusion Criteria:

* persons under the age of 18 or over the age of 75
* patients with pure receptive aphasia
* co-morbid CNS disease
* primary motor/oral apraxia
* pregnant or nursing women
* have a history of unstable mood disorder or unstable anxiety disorder or psychosis
* use of a hearing aid
* have a cochlear implant
* have a diagnosed vestibular dysfunction
* abuse alcohol or other drugs
* have had eye surgery within the previous three months or ear surgery within the previous six months
* have active ear infections or a perforated tympanic membrane
* have participated in another clinical trial within the last 30 days or are currently enrolled in another clinical trial
* Though not excluded, patients taking anti-histamines or anti-nausea drugs will be encouraged not to take such medications within four hours prior to a CVS treatment. The Investigator should review other medications taken by the patient with properties that mimic anti-nausea or anti-dizziness drugs as these may reduce responsiveness of the vestibular system to caloric stimulation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-10; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Measure and quantify any improvements in verbal fluency at the end of a 3-month Tx period | after completing 84 days of device use
  At the end of the 84 day period of device use, the patient's verbal fluency will be compared with the baseline level to assess any improvement. Boston Diagnostic Aphasia exam, Hopkins verbal learning test, oral symbol digit modality test, oral trail marking test.

SECONDARY OUTCOMES:
Mood & QoL | after completing 84 days of device use
  At the end of the 84 day period of device use, the patient's mood will be compared with the baseline scores to assess any improvement: Patient Health Questionnaire-9, Beck Depression Inventory, and for QoL: Stroke impact scale (short form), Everyday Cognition.
Gait and posture | after completing 84 days of device use
  At the end of the 84 day period of device use, the patient's gait and posture will be compared with the baseline levels to assess any improvement. This is a blended measure employing Timed Up & Go and a 10-meter walk.
Heart rate variability (HRV) | after completing 84 days of device use
  At the end of the 84 day period of device use, the patient's HRV values will be compared with those from the baseline period to assess any improvement.
Durability of gains | 3 months after the completion of therapy
  Three months after the completion of the therapy period, measurements of verbal fluency, mood & QOL, gait & posture and HRV will be completed and compared with the values from the end of the treatment period to assess durability of any gains.

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States